CLINICAL TRIAL: NCT04820569
Title: Long-term Heart-specific Mortality in the Presence of Competing Risks Among Patients With Non-metastatic Gastric Adenocarcinoma Undergoing Resection and Chemotherapy A Population-based Cohort Study of 21,257 Cases, 2004-2016
Brief Title: Long-term Heart-specific Mortality in the Presence of Competing Risks Among Patients With Non-metastatic Gastric Adenocarcinoma Undergoing Resection and Chemotherapy
Acronym: GaCCoR-01
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Lei Huang, Dr., The First Affiliated Hospital of Anhui Medical University
Other Study IDs: GaCCoR-01
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Long-term Heart-specific Mortality in the Presence of Competing Risks Among Patients With Gastric Adenocarcinoma Undergoing Resection and Chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Resection and chemotherapy

SUMMARY:
In this population-based cohort study, data on patients diagnosed with nmGaC in 2004 through 2016, managed with resection and chemotherapy, followed up until the end of 2016, and surviving ≥1 month were retrieved from the US Surveillance, Epidemiology, and End Results-18 Program. Cumulative mortality functions were calculated. Prognostic factors for heart-specific mortality were evaluated using both multivariable-adjusted Fine-Gray subdistribution and cause-specific hazard functions.

ELIGIBILITY:
Cases of non-metastatic gastric adenocarcinoma (nmGaC) were defined as patients with microscopically-confirmed first primary invasive adenocarcinoma of the stomach (International Classification of Diseases for Oncology, Third Edition (ICD-O-3) code: C16) without distant metastasis. Only those who underwent resection in January 2004 through December 2016 were included. Cancers of other histology types including squamous cell carcinoma, gastrointestinal stromal tumor or sarcoma, neuroendocrine tumor or carcinoid, lymphoma, and germ-cell tumor were ineligible, as were patients with non-gastric cancers involving the stomach, with benign or in situ tumors, or with other malignancies before gastric cancer. We further excluded patients with diagnosis based on death certificate only or autopsy, with missing follow-up period, survival status, or cause of death, or with unknown metastasis status. Cancers with distant metastasis were excluded since resection is not routinely recommended for them. Data before 2004 were not included, as the TNM stage information was unavailable. To minimize the effect of perioperative events on survival, we excluded patients surviving <1 month. No restrictions were applied to age, and patients ≥80 years only comprised 5% of those receiving both resection and chemotherapy.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases of non-metastatic gastric adenocarcinoma (nmGaC) were defined as patients with microscopically-confirmed first primary invasive adenocarcinoma of the stomach (International Classification of Diseases for Oncology, Third Edition (ICD-O-3) code: C16) without distant metastasis. Only those who underwent resection in January 2004 through December 2016 were included.
Sampling Method: Non-Probability Sample
Enrollment: 21257 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative mortality | Jan 12, 2020-Mar 5, 2021
  Cumulative incidence functions (CIFs), which, unlike the standard Kaplan-Meier method, allow for estimation of the incidence of the occurrence of an event while taking competing risks from other causes of death into account, were computed and plotted for cause-specific mortalities.
Prognostic factors for disease-specific mortalities | Jan 12, 2020-Mar 5, 2021
  Evaluated using both multivariable-adjusted Fine-Gray subdistribution and cause-specific hazard functions.

IPD SHARING:
Plan to Share IPD: Undecided
The Surveillance, Epidemiology, and End Results Program data are available upon reasonable request and with permission of the registry.